CLINICAL TRIAL: NCT05524779
Title: Evaluation of Safety and Efficacy of the BTL-785F Device for Non-invasive Reduction of Wrinkles and Overall Improvement of Appearance of the Face
Brief Title: BTL-785F Device for Non-invasive Reduction of Wrinkles and Overall Facial Improvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-785_CTUS1300
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Wrinkle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- BTL-785-7 Treatment (Experimental): Treatment of wrinkles with the BTL-785-7 applicator to the BTL-785F system.
  Interventions: Device: BTL-785-7

INTERVENTIONS:
Device: BTL-785-7 — Treatment with the BTL-785-7 applicator to the BTL-785F system.

SUMMARY:
This study will evaluate the clinical safety and the performance of the BTL-785F system equipped with the BTL-785-7 applicator for non-invasive treatment of facial wrinkles.

DETAILED DESCRIPTION:
The study is a multicenter single-arm, open-label, interventional study. The subjects will be enrolled and assigned into one experimental study arm. The subjects will be required to complete four (4) treatment visits and two follow-up visits.

At the baseline visit health status will be assessed and, if needed, additional tests will be performed. Inclusion and exclusion criteria will be verified and informed consent will be signed.

The treatment administration phase consists of four (4) treatment visits, delivered 5-10 days apart.

Safety measures will include documentation of adverse events (AE) including the subject's experience of pain or discomfort after the procedure. Occurrence of AE's will be checked immediately after the first treatment visit, prior/post to the every other procedure and at the follow-ups. Subjects will undergo two follow-up visits scheduled at 1 month and 3 months after the final treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects over 21 years of age seeking treatment for reduction of wrinkles and overall aesthetic improvement of the face
* Subjects should be able understand the investigative nature of the treatment, the possible benefits and side effects, and must sign the Informed Consent Form
* Presence of clearly visible wrinkles in the treated area when the face is relaxed as deemed appropriate by the Investigator
* Subjects willing and able to abstain from partaking in any facial treatments other than the study procedure during study participation
* Willingness to comply with study instructions, to return to the clinic for the required visits, and to have photographs of their face taken

Exclusion Criteria:

* Bacterial or viral infection, acute inflammations
* Impaired immune system
* Isotretinoin in the past 12 months
* Skin related autoimmune diseases
* Radiation therapy and chemotherapy
* Poor healing and unhealed wounds in the treatment area
* Metal implants
* Permanent implant in the treated area
* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body
* Facial dermabrasion, facial resurfacing, or deep chemical peeling in the treatment area within 3 months prior to the treatment
* Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles
* History of any type of cancer
* Active collagen diseases
* Cardiovascular diseases (such as vascular diseases, peripheral arterial disease, thrombophlebitis and thrombosis)
* Pregnancy/nursing or IVF procedure
* History of bleeding coagulopathies, use of anticoagulants
* Any active condition in the treatment area, such as sores, psoriasis, eczema, rash and rosacea
* Any surgical procedure in the treatment area within the last three months or before complete healing
* Poorly controlled endocrine disorders, such as diabetes
* Electroanalgesia without exact diagnosis of pain etiology
* Application in the area of chest, heart or over the eyes
* Serious psychopathological disorders (such as schizophrenia)
* Neurological disorders (such as multiple cerebrospinal sclerosis, epilepsy)
* Blood vessels and lymphatic vessels inflammation

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Noninvasive Treatment Of Wrinkles | 5 months
  Assess change in wrinkle severity according to the Fitzpatrick Wrinkle and Elastosis Scale. Baseline and post-treatment photographs will be evaluated. A statistically significant decrease of at least 1.0 score in the average score of Fitzpatrick Wrinkle and Elastosis Scale should be achieved.

SECONDARY OUTCOMES:
Skin Quality Assessment | 5 months
  Three evaluators will evaluate facial appearance according to the Global Aesthetic Improvement Scale (GAIS) using the photographs taken at the baseline, last therapy visit and both follow-up visits. Each evaluator will be asked to assign a score to a set of photographs. Facial appearance improvement to GAIS is considered when there is an increase in score of the scale. The baseline and post-treatment scores will be compared. If applicable, the statistical significance of obtained results will be analyzed in Microsoft Excel spreadsheet software. The level of significance (α) will be set as 5%.
Therapy Comfort | 5 months
  The 5-point Likert scale Therapy Comfort questionnaire will be used for evaluating the comfort during the treatment sessions. Pain sensation will be rated by the subjects from 0 (no pain) to 10 (worst possible pain).
Subject Satisfaction | 5 months
  The Subject Satisfaction questionnaire will be used for evaluating the satisfaction. The Subject Satisfaction Questionnaire will be given to subjects after the last treatment, at 1-month and 3-month follow-up. The answers to the questions related to the subjects' overall skin and face appearance will vary from "strongly agree" to "strongly disagree".

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Contour Medical, Gilbert, Arizona
  - Holden Timeless Beauty, San Marcos, California
  - Precision Skin Institute, Davie, Florida
  - Skin Care Physicians of Georgia, Macon, Georgia
  - Jennifer Levine MD, New York, New York

IPD SHARING:
Plan to Share IPD: No